CLINICAL TRIAL: NCT07010835
Title: A Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of YK012 in the Treatment of Moderate to Severe Systemic Lupus Erythematosus
Brief Title: Study of YK012 in Moderate to Severe Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YK012-4
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YK012 (Experimental): Phase Ib: Participants will receive four different target doses of YK012 in dose escalation stage to evaluate its safety and tolerability. Participants will receive two to three different target doses of YK012 in dose expansion stage to further evaluate its safety, tolerability and effectiveness in reducing disease activity. Phase II: Participants will receive either placebo or one to two different doses of YK012. The specific doses will be determined based on prior clinical trial results.
  Interventions: Drug: YK012

INTERVENTIONS:
Drug: YK012 — YK012 is a bispecific antibody targeting CD19 and CD3.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of YK012 in participants with Moderate to Severe Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
This clinical trial consists of Phase Ib and Phase II. Phase Ib consists of dose escalation stage and dose expansion stage. The main goal of dose escalation stage is to evaluate the safety and tolerability of YK012 in participants with Moderate to Severe Systemic Lupus Erythematosus (SLE), and the main goal of dose expansion stage is to evaluate the safety, tolerability and effectiveness in reducing disease activity of YK012 in participants with SLE. The main goal of phase II is to assess the efficacy of YK012 in participants with Moderate to Severe SLE. Pharmacokinetics, pharmacodynamics and immunogenicity of YK012 in participants are evaluated as secondary objectives in both phases.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years (inclusive) at screening, regardless of sex
* Meet the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for SLE, with a confirmed SLE diagnosis for at least 24 weeks at screening
* Positive for anti-dsDNA antibody and/or antinuclear antibody (ANA) and/or anti-Smith antibody at screening, as determined using the local laboratory's reference ranges at the study site
* Medium to high disease activity at screening, defined as: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥7
* Receiving stable background therapy at screening
* Capable of understanding and voluntarily participating in this clinical trial, having provided written informed consent, and able to comply with scheduled visits, treatments, examinations, and other study procedures.

Exclusion Criteria:

* Known allergy to monoclonal antibodies or exogenous human immunoglobulins, or hypersensitivity to the investigational drug or any of its components
* Received any anti-CD19/CD20 therapy or any B-cell depleting agents within 6 months prior to enrollment, or B-cell stimulatory factor inhibitors within 3 months or 5 half-lives prior to enrollment
* Received TNF inhibitors, interleukin receptor blockers, other small molecules or biologics within 3 months or 5 half-lives prior to enrollment
* Received intravenous immunoglobulins or plasmapheresis within 3 months prior to enrollment
* Used traditional Chinese medicines/herbal preparations for SLE treatment containing within 2 weeks prior to enrollment
* Received live or attenuated vaccines within 1 month prior to enrollment
* Has other autoimmune diseases, inflammatory joint diseases, or skin disorders (other than SLE) that may interfere with disease activity assessment
* History of malignancy within 5 years before screening, except for cured cases with no recurrence for at least 5 years, such as basal cell or squamous cell skin cancer, cervical carcinoma in situ, ductal carcinoma in situ of breast, or papillary thyroid cancer
* Clinically significant cardiovascular/cerebrovascular diseases within 6 months prior to screening
* Presence of QTcF interval prolongation on electrocardiogram (ECG)
* Presence of poorly controlled hypertension at screening
* History of non-SLE conditions requiring oral/intravenous/intramuscular/subcutaneous corticosteroid therapy (>2 weeks) within 6 months prior to enrollment
* Active tuberculosis at screening or untreated latent tuberculosis
* History of solid organ or bone marrow transplantation
* Presence of active infections
* Lupus nephritis requiring protocol-prohibited medications as assessed by the investigator
* Uncontrolled lupus crisis within 8 weeks prior to screening
* History of central nervous system (CNS) disorders
* Presence of clinically unstable or uncontrolled medical conditions at screening
* Presence of clinically significant abnormal laboratory test results
* Presence of active viral infections (e.g., hepatitis B, hepatitis C, HIV, or active syphilis)
* Had major surgery within 4 weeks prior to enrollment or planned during study;
* Participation in other interventional clinical trials within 4 weeks prior to enrollment
* Pregnant or lactating women, or individuals with pregnancy plans during the study and within a specified period after treatment who are unwilling to use effective contraception
* Other conditions deemed by investigators to preclude study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Ib dose escalation stage: Dose Limiting Toxicity (DLT) | From the first infusion of YK012 to Day 28 post first infusion
Adverse Event (AE) | From the first infusion of YK012 to the end of trial at 48 weeks
  An AE is defined as any untoward medical event that occurs after a participant receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
Severe Adverse Event (SAE) | From the first infusion of YK012 to the end of trial at 48 weeks
  An SAE refers to any untoward medical occurrence after the participant receives the IMP that results in one or more of the following: death, life-threatening event, permanent or serious disability or loss of function, hospitalization or prolongation of hospitalization, congenital abnormalities or birth defects.
Ib dose expansion stage and phase II: SRI-4 (Systemic Lupus Erythematosus Responder Index-4) response rates | From the first infusion of YK012 to the end of trial at 48 weeks

SECONDARY OUTCOMES:
Area Under the Curve (AUC0-t) of a serum concentration versus time profile | From pre-dose of YK012 to the end of trial at 48 weeks
Area under the blood concentration-time curve from zero to infinity (AUC0-∞) | From pre-dose of YK012 to the end of trial at 48 weeks
Maximum Concentration (Cmax) of YK012 | From pre-dose of YK012 to the end of trial at 48 weeks
Time to Reach Cmax (Tmax) | From pre-dose of YK012 to the end of trial at 48 weeks
Elimination Half Life (t1/2) | From pre-dose of YK012 to the end of trial at 48 weeks
Apparent Clearance (CL) | From pre-dose of YK012 to the end of trial at 48 weeks
Apparent volume of distribution (Vd) | From pre-dose of YK012 to the end of trial at 48 weeks
Minimum Concentration (Cmin) of YK012 | From pre-dose of YK012 to the end of trial at 48 weeks
Phase II: Characteristics of peripheral blood B-cell changes | From pre-dose of YK012 to the end of trial at 48 weeks
Change in urinary protein from baseline in patients with positive urinary protein during the trial | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in anti-dsDNA antibody level from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in complement C3 level from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in complement C4 level from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in IgG level from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in IgM level from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Changes in IgA levels from baseline | From pre-dose of YK012 to the end of trial at 48 weeks
Anti-Drug Antibody (ADA) positivity rate | From pre-dose of YK012 to the end of trial at 48 weeks
Neutralizing antibody (Nab) positivity rate | From pre-dose of YK012 to the end of trial at 48 weeks
Ib dose escalation stage: Systemic Lupus Erythematosus Responder Index-4 (SRI-4) response rates | From screening to the end of trial at 48 weeks
BILAG-based Composite Lupus Assessment (BICLA) response rates | From screening to the end of trial at 48 weeks
Proportion of patients achieving disease remission as defined by Definition of Remission in SLE (DORIS) | From screening to the end of trial at 48 weeks
Proportion of patients achieving Lupus Low Disease Activity State (LLDAS) | From screening to the end of trial at 48 weeks
Proportion of patients with baseline Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) score ≥10 who achieved ≥50% improvement in CLASI (CLASI-50) during the trial | From screening to the end of trial at 48 weeks
Proportion of patients with baseline ≥4 swollen and/or tender joints who achieved ≥50% improvement in joint count during the trial | From screening to the end of trial at 48 weeks
Proportion and duration of patients with baseline glucocorticoid dosage >5mg/day prednisone (or equivalent) achieving dosage ≤5mg/day prednisone (or equivalent) | From screening to the end of trial at 48 weeks
Time to relapse after achieving Lupus Low Disease Activity State (LLDAS) during the trial | From screening to the end of trial at 48 weeks
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score from baseline | From screening to the end of trial at 48 weeks
Change in British Isles Lupus Assessment Group 2004 (BILAG-2004) score from baseline | From screening to the end of trial at 48 weeks
Change in Physician's Global Assessment (PGA) score from baseline | From screening to the end of trial at 48 weeks
Change in 36-Item Short Form Health Survey (SF-36) score from baseline | From screening to the end of trial at 48 weeks
Change in Fatigue Severity Scale (FSS) score from baseline | From screening to the end of trial at 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China